CLINICAL TRIAL: NCT04498013
Title: A Clinical Study of the Effects of Cyclodynon® Compared With a Control Group on Reducing the Cumulative Risk of Breast Cancer Development in a Female Population Aged 40-52 Years With Mastodynia and BI-RADS Category 3
Brief Title: Study of the Effects of Cyclodynon on Reducing the Cumulative Risk of Breast Cancer Development in a Female Aged 40-52
Acronym: BIO-CYCL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Struk Tetiana (Other)
Collaborators: Bionorica SE (Industry)
Responsible Party: Sponsor-Investigator, Dr. Struk Tetiana, Associate professor, National University of Pharmacy
Organization: National University of Pharmacy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 453190
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Mammographic Breast Density
MeSH Terms: interventions — Vitex agnus castus extract

STUDY DESIGN:
Intervention Model Description: Female patients aged 40 to 52 years (inclusive) with mastodynia and BI-RADS category 3, who meet the requirements of inclusion/exclusion criteria will be randomized in 2 groups. The main group will be treated with Cyclodynon 1 tab per day - 6 month in addition to lifestyle modification. The control group lifestyle modification only. Dynamics of mammographic breast density (changing in BI-RADS score of category 3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Patients will be treated with Cyclodynon 1 tablet per day 6 month in addition to lifestyle modification
  Interventions: Drug: Cyclodynon; Behavioral: Lifestyl modification
- Control group (Other): Lifestyle modification only
  Interventions: Behavioral: Lifestyl modification

INTERVENTIONS:
Drug: Cyclodynon — Cyclodynon 1 tablet a day during 6 menthes period.
  Other Names: Chaste Berry (Vitex agnus-castus) Extact , 4 mg.
  Arms: Treatment group
Behavioral: Lifestyl modification — Measures to normalize the hygiene of work and rest. A diet aimed at achieving an optimal body mass index. Teaching relaxation techniques to increase resistance to chronic stress.

SUMMARY:
Increased mammographic density of mammary gland tissues and hyperprolactinaemia are regarded as one of the risk factors for the development of breast cancer in women aged 40 to 52 years, which necessitates closer monitoring of the mammary gland and can be considered as modifiable. The herbal drug Cyclodynone® has a dopaminergic effect on the hypothalamus, which causes its inhibitory effect on the secretion of prolactin. At present, a significant positive clinical and scientific experience has been accumulated in the use of the Cyclodynone® for the treatment of benign breast dysplasias against a background of mild hyperprolactinaemia in women of reproductive age. Demonstration of the positive effect of this drug on the reduction of hyperprolactinemia, mammographic density of MF, evaluation on the scale BI-RADS would justify its application for the modification of this risk factor in women aged 40 to 52 years.

DETAILED DESCRIPTION:
Hypothesis: Increased mammographic density of mammary gland tissues and hyperprolactinaemia are regarded as one of the risk factors for the development of breast cancer in women aged 40 to 52 years, which necessitates closer monitoring of the mammary gland. However, this risk factor can be considered as modifiable. The drug Cyclodynone® (contains 4 mg of special extract of dried fruits of Chaste Berry (Vitex agnus-castus)) has a dopaminergic effect on the hypothalamus, which causes its inhibitory effect on the secretion of prolactin. At present, a significant positive clinical and scientific experience has been accumulated in the use of the Cyclodynone® for the treatment of benign breast dysplasias against a background of mild hyperprolactinaemia in women of reproductive age. However, the experience of using Cyclodynone® in women older than 40-52 years with increased density or dyshormonal pathology of breast cancer is limited. Demonstration of the positive effect of this drug on the reduction of hyperprolactinemia, mammographic density of MF, evaluation on the scale BI-RADS would justify its application for the modification of this risk factor in women aged 40 to 52 years.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 40 to 52 years (inclusive) with mastodynia and BI-RADS category 3.
* The patient's written informed consent to participate in any study-related procedures.
* According to the Investigator, the patient's ability to comply with all the requirements of the study protocol, i.e. the patient's ability to cooperate adequately.
* Patients who do not have chronic diseases of the cardiovascular system, neuroendocrine system, kidneys, liver, gastrointestinal tract, respiratory system, skin in the decompensation stage.
* Consent to use reliable, evidence-based contraceptive methods (double containing the following types: hormonal, barrier, intrauterine spiral, etc.) throughout the study (from the time of the Informed Consent to Visit 6) .

Exclusion Criteria:

* Hypersensitivity to the components of the IMP.
* Burdened history of allergies.
* Participation in another clinical study less than 90 days before signing the informed consent form.
* History of cancer.
* Pregnancy or lactation.
* Administration of dopamine agonists, dopamine antagonists, oestrogens and antiestrogens, dopamine.
* Secondary amenorrhoea within 6 months or more.
* Surgical, pharmacological or physiological menopause (except hysterectomy).
* The prolactin level is more than 80 ng/mL.
* Other reasons which make the patient's participation in the study undesirable, according to the Investigator.

Ages: 40 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Research refers to the study of a pathological condition that occurs (applicable) only in the female population.
Enrollment: 150 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Mammographic density | 6 month
  Decrease in the mammographic density determined by a mammographic breast examination at Visit 5 compared to baseline (Visit 1).

SECONDARY OUTCOMES:
BI-RADS indicator | 6 month
  Dynamics of BI-RADS indicator determined by a mammographic breast examination.

CONTACTS AND LOCATIONS:
Overall Officials: Tetiana Struk, Ph.D, Principal Investigator — NFAU
Locations (1):
- Clinical and diagnostics center, Kharkiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee CI, Chen LE, Elmore JG. Risk-based Breast Cancer Screening: Implications of Breast Density. Med Clin North Am. 2017 Jul;101(4):725-741. doi: 10.1016/j.mcna.2017.03.005. PMID 28577623